CLINICAL TRIAL: NCT01097044
Title: A Phase II, Multicentre, Double-Blind, Randomised, Placebo-Controlled Study to Confirm the Safety and Efficacy of Subcutaneous Bioresorbable Afamelanotide Implants in Patients With Erythropoietic Protoporphyria (EPP)
Brief Title: Phase II Confirmatory Study in Erythropoietic Protoporphyria (EPP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CUV030
Record Dates: First submitted 2010-03-30; First posted 2010-04-01 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Erythropoietic Protoporphyria
Keywords: Erythropoietic Protoporphyria; EPP; Afamelanotide
MeSH Terms: conditions — Protoporphyria, Erythropoietic | interventions — afamelanotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Afamelanotide (Experimental): Dose: 16 mg implant; release of 16 mg over 7 to 10 days Mode of administration: Subcutaneous implantation Frequency: Every 60 days (on Days 0, 60 and 120)
  Interventions: Drug: Afamelanotide
- Placebo (Placebo Comparator): Dose: 16 mg implant; Mode of administration: Subcutaneous implantation Frequency: Every 60 days (on Days 0, 60 and 120)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Afamelanotide — One 16mg subcutaneous implant every 2 months for 6 months. (3 implants in total)
  Arms: Afamelanotide
Drug: Placebo — One placebo subcutaneous implant every 2 months for 6 months. (3 implants in total)
  Arms: Placebo

SUMMARY:
This is a randomized placebo-controlled study to be conducted in two parallel study arms for a six month period (three doses). Approximately 10 eligible patients per center will be enrolled and will receive afamelanotide (16 mg implants) or placebo according to the following dosing regimen:

* Group A will be administered afamelanotide implants on Days 0, 60 and 120
* Group B will be administered placebo implants on Days 0, 60 and 120

To determine eligibility for study inclusion, patients will undergo a screening evaluation 7 to 14 days prior to the administration of the first dose. The number and severity of phototoxic reactions will be determined Days 60, 120, and 180. Quality of life will be measured using the EPP specific questionnaire (EPP-QoL) every 60 days and the DLQI questionnaire every 7 days, beginning at Day 0 until Day 180. Participants will visit the clinic on Days 60, 120 and 180 for assessments of adverse events.

DETAILED DESCRIPTION:
Afamelanotide is a man-made drug being studied for use as a preventative medication for EPP sufferers. It is a synthetically produced analogue of human alpha melanocyte stimulating hormone (alpha-MSH) and is not yet available on the market.

The purpose of this study is to look at whether afamelanotide can reduce the number and severity of EPP symptoms when patients are exposed to light between 10:00 and 20:00 hours. This study will also look at how the drug is tolerated when taken by people with EPP.

The study will involve the use of an implant, which comes in the form of a small rod to be administered under the skin. The implant may contain the study drug afamelanotide or a placebo (inactive medication).

Over 450 subjects have been treated with afamelanotide to date with no serious safety concerns identified. For this study, afamelanotide has been formulated as a controlled release depot injection (implant). This means that the afamelanotide will be released slowly into the body over a few days. Once inserted, the implant will remain in the body after afamelanotide has been released and will slowly dissolve.

This study will help to provide more information about afamelanotide. This information will be used to determine the safety and efficacy (the ability of the drug to produce an effect) of this drug in EPP sufferers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with characteristic photosensitivity of EPP symptoms and positive diagnosis of EPP confirmed by laboratory result of elevated total protoporphyrin IX.
* Aged 18 years old and above (inclusive).
* Able to understand and sign the written Informed Consent Form.
* Willing to take precautions to prevent pregnancy until completion of the study (Day 180).

Exclusion Criteria:

* Any allergy to afamelanotide or the polymer contained in the implant or to lidocaine or other local anesthetic to be used during the administration of the study medication
* EPP patients with significant hepatic involvement
* Personal history of melanoma or dysplastic nevus syndrome.
* Current Bowen's disease, basal cell carcinoma, squamous cell carcinoma, or other malignant or premalignant skin lesions.
* Any other photodermatosis such as PLE, DLE or solar urticaria.
* Any evidence of clinically significant organ dysfunction or any clinically significant deviation from normal in the clinical or laboratory determinations.
* Acute history of drug or alcohol abuse (in the last 6 months).
* Patient assessed as not suitable for the study in the opinion of the Investigator (e.g. noncompliance history, allergic to local anesthetics, faints when given injections or giving blood).
* Participation in a clinical trial for an investigational agent within 30 days prior to the screening visit.
* Prior and concomitant therapy with medications which may interfere with the objectives of the study, including drugs that cause photosensitivity or skin pigmentation within 60 days prior to the screening visit.
* Female who is pregnant (confirmed by positive serum β-HCG pregnancy test prior to baseline) or lactating.
* Females of child-bearing potential (pre-menopausal, not surgically sterile) not using adequate contraceptive measures (i.e. oral contraceptives, diaphragm plus spermicide, intrauterine device).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Desnick, MD, Principal Investigator — Mt. Sinai
Locations (6):
- United States (6):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Mt. Sinai, New York, New York
  - Carolina's Medical Center Cannon Research, Charlotte, North Carolina
  - University of Texas, Galveston, Texas
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Recruitment period: April2010 - July2010
  Study site location:
  Mt. Sinai, New York Carolinas Medical Center, North Carolina University of Alabama at Birmingham, Alabama University of Utah, Utah University of Texas Medical Branch, Texas University of California, San Francisco, California
Period: Overall Study
Arm/Group | Afamelanotide | Placebo
Started | 39 | 38
Completed | 34 | 33
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Afamelanotide | Placebo | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (14.5) | 42.6 (15.7) | 40.3 (15.2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 0 | 3
  Between 18 and 65 years | 35 | 36 | 71
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 23 | 20 | 43
Region of Enrollment [Number; unit: participants]
  United States | 39 | 38 | 77

OUTCOME MEASURES:

1. Primary Outcome: Time in Direct Sunlight Between 10:00-15:00 on Pain-free Days
Description: The amount of direct sunlight exposure between 10:00 and 15:00 hours on days when no pain was experienced (e.g. 11-point Likert pain score of 0). Time was recorded in a patient dairy using 15 minute time blocks.
  The pain score is measured by the 11-point Likert Pain scale with minimum of 0 and maximum of 10.
  Likert Pain scale of 0 represents no pain and 10 represents worst imaginable pain.
Time Frame: Daily for 6 months
Population: One active participant and one placebo participant withdrew after Baseline assessment and no data was provided for the analysis of this endpoint.
  The overall number of participants analyzed differs from the total number of study participants because the data was either incomplete and/or missing.
Measure: Median (Full Range); unit: Hours
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 38 | 37
Hours | 8.25 [0 to 48.3] | 0.75 [0 to 71.3]

2. Secondary Outcome: Maximum Severity of Phototoxic Reaction Experienced by Participants
Description: The days on which the participant experienced pain as a result of phototoxic reactions (caused by exposure to natural light) was recorded in a study diary. On each day such a reaction occurred, the participant scored the level of pain using an 11-point Likert pain scale, with minimum of 0 and maximum of 10. The 11-point Likert pain scale with a value of 0 represents no pain and 10 represents worst imaginable pain.
  The maximum severity of a phototoxic reaction was determined by the highest daily 11-point Likert scale score that occurred during that phototoxic reaction.
Time Frame: Daily for 6 months
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 38 | 37
score on a scale | 5.0 [0 to 8] | 5.0 [0 to 10]

3. Secondary Outcome: Quality of Life Measured by Participant Completed Questionnaire
Description: Erythropoietic Protoporphyria Quality of Life Measure (EPP-QoL) is used to measure the quality of life of participants.
  The total EPP-QoL score ranges from 0 to 100, with a score of 0 as the worst quality of life and score of 100 as the best quality of life.
Time Frame: Day 0, Day 60, Day 120, Day 180
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 38 | 37
units on a scale
  Day 0 | 34.7 [3 to 67] | 22.2 [3 to 78]
  Day 60: number analyzed (Participants) | 38 | 35
  Day 60 | 73.6 [17 to 100] | 44.4 [6 to 94]
  Day 120: number analyzed (Participants) | 36 | 34
  Day 120 | 84.7 [6 to 100] | 55.6 [6 to 100]
  Day 180: number analyzed (Participants) | 34 | 35
  Day 180 | 88.9 [56 to 100] | 63.9 [0 to 100]

4. Secondary Outcome: Change of Total Protoporphyrin IX Level in Participants
Description: This was an exploratory assessment only to analyze whether afamelanotide-induced change in sun exposure would result in a reduction of protoporphyrin IX.
  The changes of the Total Protoporphyrin IX Level (μg/dL) from Screening Visit (ITT Population) were measured between the two groups.
  The Protoporphyrin IX level is a laboratory parameter that is measured in specialist labs.
Time Frame: Baseline, Day 60, Day 120, Day 180
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 38 | 37
mcg/dL
  Day 60: number analyzed (Participants) | 38 | 35
  Day 60 | -471.3 (505.4) | -628.5 (837.5)
  Day 120: number analyzed (Participants) | 36 | 34
  Day 120 | -511.8 (595.3) | -619.9 (1022.3)
  Day 180: number analyzed (Participants) | 34 | 37
  Day 180 | -92.7 (549.1) | -369.2 (1265.6)

5. Secondary Outcome: Number of Participants With Phototoxic Reactions With Likert Severity Scores ≥ 4 and ≥ 7
Description: The number of participants who experienced phototoxic reactions with Likert severity scores ≥ 4 and severity scores ≥7 were recorded.
  A derived endpoint was used. The number of participants who reported at least one phototoxic reaction with a Likert severity score of ≥ 4 was recorded. For severity scores ≥ 7, the number of patients who reported at least one phototoxic reaction with a Likert severity score of ≥ 7 was recorded.
  The 11-point Likert pain scale ranges from minimum of 0 to maximum of 10. The 11-point Likert pain scale with a value of 0 represents no pain and 10 represents worst imaginable pain.
Time Frame: Daily for 6 months
Population: as for outcome 1
Measure: Number; unit: Count of Participants
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 38 | 37
Count of Participants
  Severity Likert score of ≥ 4 | 26 | 24
  Severity Likert score of ≥ 7 | 7 | 14

6. Secondary Outcome: Number of Phototoxic Reactions Experienced by Participants
Description: The days on which the participant experienced pain as a result of phototoxic reactions (caused by exposure to natural light) was recorded in a study diary. On each day such a reaction occurred, the participant scored the level of pain using an 11-point Likert pain scale, with minimum of 0 and maximum of 10. The 11-point Likert pain scale with a value of 0 represents no pain and 10 represents worst imaginable pain.
  The number of phototoxic reactions was determined by counting the number of episodes on which participants report a 11-point Likert scale score of 4 or more for one or more consecutive days.
Time Frame: Daily for 6 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Episodes
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 38 | 37
Episodes | 2.0 [0 to 25] | 1.0 [0 to 13]

7. Secondary Outcome: Total Severity of Phototoxic Reactions Experienced by Participants Over the Entire Study
Description: The days on which the participant experienced pain as a result of phototoxic reactions (caused by exposure to natural light) was recorded in a study diary.
  On each day such a reaction occurred, the participant scored the level of pain using an 11-point Likert pain scale, with minimum of 0 and maximum of 10. The 11-point Likert Pain scale with a value of 0 represents no pain and 10 represents worst imaginable pain.
  The total severity of phototoxic reactions was determined by the sum of daily 11-point Likert scale scores that occurred during phototoxic reactions. The overall sum of the severity per participant over the entire study was analyzed. The theoretical minimum score is 0 and the maximum possible score is 1800.
Time Frame: Daily for 6 months.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 38 | 37
units on a scale | 27.9 (43.1) | 37.2 (102.6)

ADVERSE EVENTS:
Time Frame: 6 months (180 days)
Arm/Group | Afamelanotide | Placebo
Serious Adverse Events (participants affected / at risk) | 2/39 | 2/38
Other Adverse Events (participants affected / at risk) | 31/39 | 29/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afamelanotide (N=39) | Placebo (N=38)
CRAMPY ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 1
Low Pulse Rate (Cardiac disorders) | 0 | 1
RECURRENT RECTAL BLEEDING (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afamelanotide (N=39) | Placebo (N=38)
Nausea (Gastrointestinal disorders) | 8 | 2
Abdominal discomfort (Gastrointestinal disorders) | 3 | 2
Fatigue (General disorders) | 3 | 1
Implant Site Pain (General disorders) | 1 | 5
Pyrexia (General disorders) | 3 | 1
Nasopharyngitis (Infections and infestations) | 7 | 2
Sinusitis (Infections and infestations) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Headache (Nervous system disorders) | 5 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No